CLINICAL TRIAL: NCT06623448
Title: Nursing Students&Amp;#39; Readiness for Medical Artificial Intelligence and Artificial Intelligence Anxiety: A Mixed Method Study
Brief Title: Nursing Students and Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Rukiye Burucu, Assistant Prof, Necmettin Erbakan University
Other Study IDs: Artificial Intelligence
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Nursing Students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nursing students

SUMMARY:
The aim of this observational study is to examine nursing students' readiness for medical AI and their anxiety about AI using a mixed method.

The main question it aims to answer is:

Nursing students';

1. What is their level of awareness of medical artificial intelligence?
2. What is their level of artificial intelligence anxiety?
3. Is there a relationship between artificial intelligence awareness and anxiety levels?
4. What are the opinions of those who have artificial intelligence anxiety about artificial intelligence?

In the 1st stage, nursing students answered the related survey questions online. In the 2nd stage, qualitative interviews were conducted with those with high AI anxiety scores and evaluated.

ELIGIBILITY:
Inclusion Criteria:

To be a student of Necmettin Erbakan University Faculty of Nursing To be a student of Necmettin Erbakan University Kamil Akkanat Faculty of Health Sciences, Department of Nursing

Exclusion Criteria:

Students who did not consent to participate were excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 977
Sampling Method: Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Artificial intelligence awareness level and artificial intelligence anxiety leve | Until the end of August 2025
  Mean score of medical artificial intelligence awareness scale and mean artificial intelligence anxiety scale score

SECONDARY OUTCOMES:
Students' views on artificial intelligence | 5th September
  Students' views will be obtained through a focus group interview

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Still undecided

REFERENCES:
- [Derived] Burucu R, Turkben Polat H. Nursing students' readiness and anxiety regarding medical artificial intelligence: A mixed-methods study. Nurse Educ Pract. 2025 Oct;88:104538. doi: 10.1016/j.nepr.2025.104538. Epub 2025 Sep 9. PMID 40957231